CLINICAL TRIAL: NCT06382792
Title: Results of Proximal Humeral Reconstruction With Allograft Prosthetic Composite After Resection for Tumors
Brief Title: Osteolysis of Allograft Prosthetic Composite After Shoulder Resection for Tumors
Status: Enrolling by invitation | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, PEDUZZI Lisa, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2024PI059
Record Dates: First submitted 2024-04-15; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Shoulder Disease
MeSH Terms: interventions — Tumor Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: proximal humeral resection for tumor and allograft prosthetic composite reconstruction — allograft prosthetic composite

SUMMARY:
The gold standard after shoulder resection for tumors is reconstruction by reverse prosthesis and allograft. This is an intervention also performed for more frequent etiologies (revisions of prosthesis, non cancerous humeral bone loss ...).

The results in these etiologies are good, and do not find any particular mechanical complications (including no osteolysis of the graft). In the case of reconstruction for cancer, the numbers of patients are lower (rare pathologies) and some studies on small numbers found osteolysis of the allograft. The aim of this study is to analyze the presence or not osteolysis in these patients, and to quantify it precisely by scanner measurement (no data yet in the literature).

DETAILED DESCRIPTION:
quantify bone stock of the allograft by scanner measurement in post operative and in 6 month to 1 years after surgery.

This is a retrospective study, and the scanner was performed routinely every 3 to 6 month, during 2 years, for oncological follow up.

ELIGIBILITY:
Inclusion Criteria:

* tumors of proximal humerus
* Malawer type I resection
* primary reconstruction by allograft prosthetic composite

Exclusion Criteria:

* resection and reconstruction by prosthesis alone
* resection and reconstruction by prosthesis and cement sleeve reconstruction
* resection and reconstruction by hemiarthroplasty
* revision protheses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated for tumors of proximal humerus, who underwent a Malawer type I resection of this tumors
Sampling Method: Non-Probability Sample
Enrollment: 6 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Osteolysis (bone stock in cm3) | within 3 months post operatively and up to 1 year post operatively
  allograft bone stock by scanographic measurements after the surgery, and at minimum 6 month follow up

SECONDARY OUTCOMES:
Constant score | up to 1year post operatively
  Shoulder functional evaluation score between 6 points (worst score) and 100 points (better score)
Complications | up to 1year post operatively
  (infection, dislocation)
Revision | up to 1year post operatively
  with removal of implant, with or without re implantation

CONTACTS AND LOCATIONS:
Overall Officials: Sirveaux FRANCOIS, Study Chair — Central Hopital, Nancy France
Locations (1):
- Central Hopital, Nancy, France

IPD SHARING:
Plan to Share IPD: No